CLINICAL TRIAL: NCT04979572
Title: A Phase 1, Single-Center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending and Multiple Dose of TS-172 in Healthy Adult Subjects
Brief Title: A Phase I Study of TS-172 in Healthy Adult Subjects (Single and Multiple Doses)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TS172-101
Record Dates: First submitted 2021-07-05; First posted 2021-07-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (single dose) : Step 1 to 4: TS-172 10 mg, 30 mg, 90 mg, 270 mg (Experimental): Single dose of TS-172 or placebo before breakfast
  Interventions: Drug: TS-172; Drug: Placebo
- Part B (multiple dose) : Step 5: TS-172 90 mg (Experimental): Multiple dose of TS-172 or placebo before breakfast and dinner
  Interventions: Drug: TS-172; Drug: Placebo

INTERVENTIONS:
Drug: TS-172 — * Single doses of TS-172 10 mg, 30 mg, 90 mg, 270 mg before breakfast in each period (only 30 mg administered before breakfast and fasting)
  * Multiple dose of TS-172 90 mg before breakfast and dinner
Drug: Placebo — * Single doses of TS-172 placebo before breakfast in each period (only placebo administered before breakfast and fasting in step 2)
  * Multiple dose of TS-172 placebo before breakfast and dinner

SUMMARY:
A Phase 1, Single-Center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending and Multiple Dose of TS-172 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Japanese healthy males aged 20 years or older but less than 40 years at the time of informed consent
2. Those with a BMI of 18.5 or more and less than 25.0 at screening test
3. Those who are able to receive the explanation before participating in the study, understand the content of the study, and provide written informed consent by the subjects themselves.

Exclusion Criteria:

1. Subjects who have any disease and are not considered healthy subjects based on the medical judgment of the principal investigator or sub-investigator.
2. Those who correspond to any of the following about bowel movements;

   * Repeated diarrhea (Bristol Stool Form Score [BSFS] score of 6 or higher) on a daily basis
   * Repeated constipation (no defecation for 2 days or more in a week) on a daily basis
3. Those who correspond to any of the following about bowel movements in the 7 days before administration;

   * Diarrhea on 2 or more days in 7 days
   * 2 or more days without a bowel movement in 7 days
4. Those who have a history of gastrointestinal ulceration
5. Those who correspond to any of the following about infection;

   * Positive for SARS-CoV-2 in the nucleic acid amplification test performed at the time of admission
   * Suspected of having COVID-19

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious AEs (SAEs) | Part A (Step 1): Day 1 up to Day 8, Part A (Step 2, 3, 4): Day 1 up to Day 4, Part B: Day 1 up to Day 11

SECONDARY OUTCOMES:
Concentration of unchanged form in plasma, urine and stool | Part A: Day 1 up to Day 4, Part B: Day 1 up to Day 11
Area under the plasma concentration-time curve (AUC) of unchanged form | Part A: Day 1 up to Day 4, Part B: Day 1 up to Day 11
Mean daily urinaly excretion of sodium and phosphorus | Part A (Step 1): Day 1 up to Day 8, Part A (Step 2, 3, 4): Day 1 up to Day 4, Part B: Day 1 up to Day 11
Mean daily Bristol Stool Form Scale (BSFS) | Part A (Step 1): Day 1 up to Day 8, Part A (Step 2, 3, 4): Day 1 up to Day 4, Part B: Day 1 up to Day 11
  BSFS is a scale between 1-7, where 1 correlates with the firmest stool and 7 correlates with entirely liquid stool

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Toshima-ku, Japan

IPD SHARING:
Plan to Share IPD: No